CLINICAL TRIAL: NCT05703529
Title: The Impact of Group-based Positive Psychotherapy in Psychological Resilience of Only-child-lost People: A Randomized Controlled Trial
Brief Title: Group-based Positive Psychotherapy in Psychological Resilience of Only-Child-Lost People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Zhang Wen, Xiangya School of Nursing, Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015058
Record Dates: First submitted 2022-12-20; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Resilience, Psychological; Bereavement; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention provider, investigator, and outcomes assessor have not been informed of the group allocation, but the participants may be aware of the group allocation because of the nature of the research design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychotherapy group (Experimental)
  Interventions: Behavioral: Positive Psychotherapy
- Control group (Other): Usual Care means treating as usual, including a regular home visit.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Positive Psychotherapy — A 6-week group-based positive psychotherapy was conducted in this group. The themes of each week include positive introduction, three good things and positive reactions, gratitude, positive memory, identifying personal strengths and utilizing strengths.
  Arms: Positive Psychotherapy group
Other: Usual Care — Usual Care means treating as usual, including a regular home visit.
  Arms: Control group

SUMMARY:
A randomized controlled trial was conducted to evaluate the effectiveness of group-based positive psychotherapy on psychological resilience, depression, well-being, sleep quality, dehydroepiandrosterone in only-child-lost people. A total of 80 only-child-lost people who met the inclusion and exclusion criteria were expected to recruit. There were six weeks in the intervention, including positive introduction, positive reaction, gratitude, meaningful, three good things, and using personal strength. The measurements were conducted at the baseline, immediately after the intervention, 3-month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. having only one child or legally adopting;
2. No surviving children;
3. basic language expression and comprehension skills;
4. the score of Connor-Davidson Resilience Scale is lower than 82

Exclusion Criteria:

1. in the acute bereavement period (<6 months);
2. unable to participate in activities due to severe physical illness;
3. having diagnosis of sever mental illness;
4. receiving other psychological therapy.

Min Age: 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Change of psychological resilience | Baseline, immediately after the intervention, 3-month after the intervention
  It is assessed by Connor-Davidson Resilience Scale. A higher score suggests a higher level of psychological resilience. The range is 0-100.

SECONDARY OUTCOMES:
Change of depressive symptoms | Baseline, immediately after the intervention, 3-month after the intervention
  It is measured by Zung Self-rating Depression Scale with a higher score suggesting a more severe of depressive symptoms
Change of index of well-being | Baseline, immediately after the intervention, 3-month after the intervention
  It is measured by Campbell's Index of Well-being. A high score indicates a high level of well-being.
Change of Dehydroepiandrosterone (DHEA) in saliva | Baseline, immediately after the intervention, 3-month after the intervention
  Saliva is collected using a saliva collector and assayed using the Elisa assay. After the specimens were collected, they were tested with the Elisa kit of Salimetrics® according to its instructions.
Change of Sleep Quality | Baseline, immediately after the intervention, 3-month after the intervention
  It is measured by Pittsburgh Sleep Quality Index. If the total score is over 7, the sleep quality is normal, and if the score is over 7, it suggests a low sleep quality
Change of Social Avoidance and Social Distress | Baseline, immediately after the intervention, 3-month after the intervention
  It is measured by Social Avoidance and Distress Scale. A high score indicates a high level of social avoidance and social distress.